CLINICAL TRIAL: NCT03798951
Title: Evaluation of a Multimodal Program of Prehabilitation in Patients Undergoing Esophagectomy Within an ERAS Pathway
Brief Title: Prehabilitation in Esophageal Surgery (PRESS)
Acronym: PRESS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated prematurely due to slow recruitment.
Sponsor: Università Vita-Salute San Raffaele (Other)
Collaborators: Stefano Turi (Unknown); Luigi Beretta (Unknown); Paolo Parise (Unknown); Riccardo Rosati (Unknown)
Responsible Party: Principal Investigator, Giovanni Landoni, MD, Asociate Professor, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRESS 152/INT/2018
Record Dates: First submitted 2019-01-07; First posted 2019-01-10 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Esophageal Cancer Surgery
Keywords: Esophageal cancer surgery; Prehabilitation; Enhanced recovery after surgery
MeSH Terms: interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation program (Experimental): The patients included in the treatment group will follow a prehabilitation program, based on a physiotherapist, nutritionist and psychologist evaluation. All the treatments will be tailored according the characteristics of each single patient. The program will have a duration of, at least, 4 weeks.
  Interventions: Other: Prehabilitation
- Control (No Intervention): The patients included in this group will, also, receive a basal evaluation by a physiotherapist, a nutritionist and a psychologist. These patients will not receive a tailored prehabilitation program and will be revaluated the day before surgery.

INTERVENTIONS:
Other: Prehabilitation — The patients included in the treatment group will follow a prehabilitation program, based on a physiotherapist, nutritionist and psychologist evaluation. All the treatments will be tailored according the characteristics of each single patient.
  The program will have a duration of, at least, 4 weeks.
  Arms: Prehabilitation program

SUMMARY:
Despite important clinical improvements, esophageal cancer surgery is still associated to a high rate of postoperative complications. Recent ERAS (Enhanced Recovery After Surgery) Society guidelines underline the possible role of prehabilitations' programs in reducing postoperative morbidity. In this trial, 200 patients, scheduled for esophageal cancer resection, will be randomly assigned to two groups (100 patients for each group). In both groups, patients will perform a basal evaluation with a physiotherapist, a nutritionist and a psychologist. In the treatment group, each patient will receive a tailored prehabilitative program and, during the 4 weeks before surgery, will be monitored constantly by each single specialist. A preoperative revaluation (the day before surgery) and follow up visits at 3 and 6 months will be performed for all patients. The incidence of postoperative complications, the length of hospital stay, and the reach of discharge criteria will be registered.

DETAILED DESCRIPTION:
Multi-modal prehabilitation programs reported positive results in patients undergoing colonic resection. These protocols are, generally, based on physiotherapist, nutritional and psychological implementation programs. Nevertheless, the conflicting results obtained in previous trials demonstrate how many elements have still to be clarified and that, probably, the pre-habilitation interventions must be tailored, as much as possible, on the peculiar characteristics of each single patient, modifying the approach as a function of the clinical specific response. All these considerations suggest a strong basis for tailored interventions in patients undergoing esophageal surgery, highlighting at the same time, as concluded in a recent review, the need of further studies to better define specific peri-operative strategies. This study will be a randomized, not blind, monocentric trial, that will be conducted at Ospedale San Raffaele, Milano, Italia, between January 2018 and January 2021 (three years). 200 patients will be randomly assigned to two different groups. All the patients, included in the study, will receive a preliminary evaluation performed by different professional figures.

Physiotherapist evaluation:

All the patients of both groups will be classified according to specific tests in order to establish their basal condition. Spirometry examination, 6-minute walking test, time up and go test, steep ramp test

strength tests (target muscles will be the quadriceps and the handgrip muscles:

in both cases a specific dynamometer will be utilized) and Modified Iowa Level

of Assistance Scale (MILAS) evaluation will be performed.

The experimental group will follow a home-based prehabilitation program for four weeks; this will be tailored on the patient on the bases of the first functional evaluation and the identified needs. On day 1 the patients will attend a hospital session and will be instructed by a physiotherapist on exercises and program to follow. The patients will then receive instruction support in order to better follow and adjust the program at home. Patients will also record what they do on a diary.

The physiotherapist will make phone calls in order to supervise patients' adherence to the program and help them in adjusting it.

Prehabilitation program will comprise aerobic exercise (cyclette or treadmill, 3 times a week) and IMT (inspiration muscle training, IMT respironics Philips, daily). In adjunction to these ones, further exercises will be prescribed on the bases of the functional assessment and the identification of deficits in any functional capacity assessed and will include two of the following: airway clearance (two sessions 10' a day for 7 days a week), skeletal muscles strengthening (3 days a week), stretching (three times a week), transfer and mobility training.

The control group will follow the actual procedure usually administered prior to surgery: this comprises inspiration exercises through a spirometer incentive without any monitoring and some recommendations aimed at staying active during the preoperative period.

Nutritional evaluation:

All patients will undergo a comprehensive nutritional assessment at baseline, 4 weeks prior to surgery, the day before or the day of surgery and 3 and 6 months after surgery. At baseline, a complete medical and nutrition history will be collected, and physical examination will be performed. Anthropometric parameters including body weight (kg) and height (cm), waist and hip circumference will be measured, and body mass index (kg/m2) calculated. The Malnutrition Universal Screening Tool (MUST) will be used to screen patients for nutrition risk. Standard biochemical markers of malnutrition and inflammation, including albumin, prealbumin, retinol-binding protein, total lymphocyte count, transferrin and C-reactive protein will be measured in all patients. The Prognostic Nutritional Index (PNI) will also be calculated using serum albumin concentration and total lymphocyte count. Single frequency-bio-impedance analysis (SF-BIA) will be used to estimate total body water (TBW), fat free mass (FFM) and BIA-derived phase angle. Basal energy expenditure (BEE) will be estimated using the Harris-Benedict equation. Energy and protein needs (ranging from 1 to 1.5 g/kg/day) will be established according to age, BEE, disease and degree of protein depletion. At baseline, all patients will receive nutrition counselling to help manage symptoms and encourage the intake of energy-enriched foods and fluids that are better tolerated, as per the European Society for Clinical Nutrition and Metabolism (ESPEN) guidelines on nutrition in cancer patients. Patients in the treatment group will be provided with a dietary plan based on their energy and protein needs. Patients will be monitored by a follow-up phone call at two weeks after the baseline visit. Furthermore, patients in the treatment group will receive an immune-enhancing formula (7.6% protein, 18.9% carbohydrate, 3.9% fat) enriched with arginine, RNA, ω3 fatty acids and soluble fibre (partially hydrolysed guar gum, PHGG) 5 days before surgery (237 ml TID). Patients in the control group will receive nutritional counselling at baseline and will be managed according to standard protocols in use at our Institution.

Psychologist evaluation:

All the patients will perform a psychological interview and specific assessment tests to define their: quality of life (SF-36 and EORTC), specific disorders anxiety and depression Hads (Hospital anxiety and Depression Scale) and coping strategies (MAC mental Adjustment to Cancer). The assessment test will be performed at the recruitment of the patients, the day before surgery and 3 and 6 months after surgery. In the treatment group, periodical re-evaluations, trough phone calls, will be performed to support patients in their adjustment path to surgery. It will be, also, necessary to sustain them to accept possible changes and pressures deriving from prehabilitative programs. Treated patients will also receive a post-operative evaluation to define possible symptoms and adaptive reactions, developed to overcome the physiologic and metabolic modifications deriving from surgery.

The intra and post-operative treatment will be developed according to the same principles of ERAS in both groups. The authors will record all post-operative complications; the length of hospital stays and the reach of the criteria for the discharge (free solid intake, adequate pain control with oral analgesics, autonomous mobilization, restarting of bowel function and no evidence of possible post-surgical complications). Postoperative complications will be defined and registered according Calvien- Dindo classification criteria. The primary outcome of our study will be the reduction of post-operative complications, from 70% to 50%. Secondary outcomes will be a reduction in the length of hospital stay and a faster return to the pre-operative physical conditions, through a comparison with the basal evaluation, in the treatment group. Patients will be evaluated the day before surgery, during hospital stay and trough a follow-up visit at 3 and 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent;
* Patients scheduled for Esophageal cancer resection with Ivor-lewis technique;
* Previous CT/RT neoadjuvant treatment;
* Possibility to perform a prehabilitation treatment of, at least, 4 weeks.

Exclusion Criteria:

* Patient refusal
* Comorbid medical, physical, and mental conditions that contraindicate exercise or oral nutrition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Post-operative complications | Hospital discharge (10-15 days)
  Reduction of incidence of post-operative complications, registered according to Clavien-Dindo's Classification criteria

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele Scientific Institute, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Low DE, Allum W, De Manzoni G, Ferri L, Immanuel A, Kuppusamy M, Law S, Lindblad M, Maynard N, Neal J, Pramesh CS, Scott M, Mark Smithers B, Addor V, Ljungqvist O. Guidelines for Perioperative Care in Esophagectomy: Enhanced Recovery After Surgery (ERAS(R)) Society Recommendations. World J Surg. 2019 Feb;43(2):299-330. doi: 10.1007/s00268-018-4786-4. PMID 30276441
- [Background] Minnella EM, Awasthi R, Loiselle SE, Agnihotram RV, Ferri LE, Carli F. Effect of Exercise and Nutrition Prehabilitation on Functional Capacity in Esophagogastric Cancer Surgery: A Randomized Clinical Trial. JAMA Surg. 2018 Dec 1;153(12):1081-1089. doi: 10.1001/jamasurg.2018.1645. PMID 30193337
- [Background] Minnella EM, Carli F. Prehabilitation and functional recovery for colorectal cancer patients. Eur J Surg Oncol. 2018 Jul;44(7):919-926. doi: 10.1016/j.ejso.2018.04.016. Epub 2018 Apr 30. PMID 29754828
- [Background] Stratton RJ, Hackston A, Longmore D, Dixon R, Price S, Stroud M, King C, Elia M. Malnutrition in hospital outpatients and inpatients: prevalence, concurrent validity and ease of use of the 'malnutrition universal screening tool' ('MUST') for adults. Br J Nutr. 2004 Nov;92(5):799-808. doi: 10.1079/bjn20041258. PMID 15533269
- [Background] Mohri Y, Inoue Y, Tanaka K, Hiro J, Uchida K, Kusunoki M. Prognostic nutritional index predicts postoperative outcome in colorectal cancer. World J Surg. 2013 Nov;37(11):2688-92. doi: 10.1007/s00268-013-2156-9. PMID 23884382
- [Background] Arends J, Bachmann P, Baracos V, Barthelemy N, Bertz H, Bozzetti F, Fearon K, Hutterer E, Isenring E, Kaasa S, Krznaric Z, Laird B, Larsson M, Laviano A, Muhlebach S, Muscaritoli M, Oldervoll L, Ravasco P, Solheim T, Strasser F, de van der Schueren M, Preiser JC. ESPEN guidelines on nutrition in cancer patients. Clin Nutr. 2017 Feb;36(1):11-48. doi: 10.1016/j.clnu.2016.07.015. Epub 2016 Aug 6. PMID 27637832